CLINICAL TRIAL: NCT06795425
Title: A Randomized, Double-Blinded, Placebo-Controlled, Parallel Study, to Assess the Effect of a Novel Postbiotic Blend on Exercise Induced Oxidative Stress Markers and Exercise Performance
Brief Title: A Randomized, Double-Blind Study to Assess the Effect of a Postbiotic on Oxidative Stress and Exercise Performance
Acronym: PBE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Collaborators: Archer Daniels Midland Co. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTB2022TN206; IRB-24-16 (Other: Lindenwood University Institutional Review Board)
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Oxidative Stress; Healthy; Exercise-induced Muscle Damage; Exercise-induced Muscle Soreness; Immune Function; Gut Health; Microbiome Analysis; Exercise Performance; Exercise Metabolism
Keywords: oxidative stress; antioxidants; postbiotics; ergogenic aid; exercise performance; muscle damage; recovery; gut microbiome; immune function; sleep quality; anxiety; recreationally active; inflammation; endurance training; fecal microbiota; nutritional supplement; aerobic exercise; biomarkers; clinical trial
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Inflammation

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, double-blind, parallel design with two groups. Participants are assigned to either the active postbiotic blend group or a placebo group to evaluate the blend's effects on oxidative stress, muscle recovery, immune function, and exercise performance.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: To maintain blinding, each participant is assigned a unique randomization number, rather than a direct treatment label (e.g., "A" or "B"). Treatments are provided with coded labels, ensuring that participants, investigators, outcome assessors, and any other study staff involved in data collection remain unaware of the group assignments throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Postbiotic Active Lifestyle Blend (Experimental): Participants in this arm will receive the active Postbiotic Active Lifestyle Blend supplement, which contains a heat-treated blend of bacterial strains
  Interventions: Dietary Supplement: Postbiotic Active Lifestyle Blend
- Placebo (Placebo Comparator): Participants in this arm will receive a placebo capsule that matches the appearance and dosage of the active blend.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Postbiotic Active Lifestyle Blend — The active intervention, Postbiotic Active Lifestyle Blend, containing a heat-treated blend of bacterial strains; 2 capsules per day.
  Arms: Postbiotic Active Lifestyle Blend
Other: Placebo — The placebo intervention contains no active ingredients and consists of maltodextrin as an inactive ingredient. The capsule matches the appearance and dosage form of the active intervention.
  Arms: Placebo

SUMMARY:
This is a prospective, randomized, placebo controlled, double-blind study to assess the effects of a postbiotic blend on exercise induced oxidative stress markers and exercise performance in healthy adult.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled study will evaluate the effect of a novel postbiotic blend on oxidative stress markers and exercise performance in healthy, physically active adults. The study aims to determine whether the postbiotic supplement can reduce oxidative stress and enhance exercise outcomes over an 8-week period.

Participants will be randomly assigned to receive either the postbiotic blend or a placebo in a double-blind fashion. The study includes an 8-week intervention period, with baseline and follow-up assessments conducted to evaluate changes in key biomarkers and performance metrics.

The primary outcome measure will focus on changes in malondialdehyde concentrations, a key marker of oxidative stress. Secondary outcomes will include assessments of other oxidative stress markers, immune function, and exercise performance. Detailed descriptions of these outcome measures are provided in the "Outcome Measures" section.

Participants will undergo a series of assessments at baseline, mid-study, and post-intervention. These assessments include blood draws, VO2 peak testing, and exercise performance tests. Participants will also be required to maintain a daily diary documenting their health status, medication/supplement use, and any adverse events.

The total study duration is 8-10 weeks, including a pre-study screening phase, 8 weeks of intervention, and a follow-up assessment.

ELIGIBILITY:
INCLUSION CRITERIA

To be eligible for inclusion, the participant must fulfill all of the following criteria:

1. Male or female participants between 18 - 45 years of age
2. Signed informed consent.
3. Health, which is defined as currently not being treated for an active cardiac, pulmonary, metabolic, immunological, neurological, respiratory, orthopedic, musculoskeletal, psychiatric, or reproductive disease or disorder. With research team and principal investigator discretion, some ongoing treatments will be permitted if a determination is made that the treatment will not increase risk of study participation and the treatment or illness itself will not confound with desired study outcomes.
4. Physically active, which is defined as performing aerobic or resistance-based physical exercise between 2 and 5 times per week at a rating of perceived intensity (RPE) of 4 or greater (out of 10)
5. Body mass index values will range from >18.5 to < 29.9 kg/m2 (Inclusive)41 (Weir and Jan 2024).
6. Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, and carry out all study-related procedures.

EXCLUSION CRITERIA

Participants will be excluded from the study if they meet any of the following criteria:

1. Body mass index <18.5 to <29.9 kg/m2 (Inclusive)
2. Use of antibiotics or probiotics in the previous 3 months
3. Positive medical history and/or is currently being treated for some form of heart or cardiovascular, neurological impairment, disease or condition, immune disorder or disease, thyroid disease, kidney disease, renal failure, regular dialysis, liver disease or other diagnosed hepatic impairment.
4. Diagnosed with having Type I or Type II diabetes (determined as fasting blood glucose > 126 mg/dL)
5. Diagnosed with major affective disorder or other significant psychiatric disorder or disturbance that required hospitalization or home intervention in the prior year.
6. History of cancer (except localized skin cancer without metastases or in situ cervical cancer within 5 years prior to screening visit).
7. Participant has an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g., dysphagia) and digestion (e.g., known intestinal malabsorption, bile acid malabsorption, H.pylori infection, small intestine bacterial overgrowth (SIBO), celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea)
8. Recently prescribed or change in dosage (within the past 6 months) of statin drug (i.e., Lipitor, Livalo, Crestor, Zocor, etc.), hypertension medications (i.e., Beta-blockers, ACE Inhibitors, Alpha blockers, Vasodilators, etc.), or psychiatric medications.
9. Consumption (any dose or amount) of any nicotine-containing product (cigarette, cigar, vaping, etc.)
10. Participants who are lactating, pregnant or planning to become pregnant.
11. History of alcohol or substance abuse in the 12 months prior to screening
12. Receipt or use of an investigational product in another research study within 60 days of beginning the study protocol.
13. Any condition or abnormality that, in the opinion of the investigator, would compromise the safety of the participant or the quality of the study data.
14. Extensive travel (>1 month) that will disrupt original outline of the study protocol.
15. Participant is consuming a biotic product (pre-, pro-, syn-, or post-) or alters their diet resulting in a change in the amount of prebiotic, probiotic, or fermented foods that are consumed while in the study protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Serum Malondialdehyde Concentrations 30 Minutes Before and 30 Minutes After Exercise Completion After 0 and 8 Weeks of Supplementation | 30 minutes before and 30 minutes after exercise completion at baseline (0 weeks) and after 8 weeks of supplementation.
  Serum malondialdehyde (MDA) concentration will be measured to assess the effect of the postbiotic blend on lipid peroxidation and oxidative stress. Higher MDA levels indicate increased oxidative stress.

SECONDARY OUTCOMES:
Change from Baseline in Urine 8-OHdG During the 24 Hours Before and 24 Hours After Exercise Completion at 0 and 8 Weeks of Supplementation | 24 hours before and 24 hours after exercise completion at baseline and after 8 weeks of supplementation.
  Urinary 8-OHdG, a biomarker for oxidative DNA damage, will be measured to evaluate oxidative stress. Values reflect the total oxidative stress experienced by participants.
Change from Baseline in Serum Oxidized LDL Concentrations 30 Minutes Before and 30 Minutes After Exercise Completion at 0 and 8 Weeks of Supplementation | 30 minutes before and 30 minutes after exercise completion at baseline and after 8 weeks of supplementation.
  Serum oxidized LDL will be measured as an indicator of oxidative modification in lipids, associated with cardiovascular risk. Higher levels represent increased lipid oxidation.
Change from Baseline in Serum Glutathione Peroxidase Activity 30 Minutes Before and 30 Minutes After Exercise Completion at 0 and 8 Weeks of Supplementation | 30 minutes before and 30 minutes after exercise completion at baseline and after 8 weeks of supplementation.
  Glutathione peroxidase levels, a measure of antioxidant enzyme activity, will be assessed in serum. Higher activity indicates greater antioxidant defense.
Change from Baseline in Urinary 8-Isoprostane Levels During the 24 Hours Before and 24 Hours After Exercise Completion at 0 and 8 Weeks of Supplementation | 24 hours before and 24 hours after exercise completion at baseline and after 8 weeks of supplementation.
  Urinary 8-isoprostane, a marker for lipid peroxidation, will be measured to assess oxidative stress. Higher values indicate greater oxidative damage to lipids.
Change from Baseline in Serum Total Antioxidant Status (TAS) 30 Minutes Before and 30 Minutes After Exercise Completion at 0 and 8 Weeks of Supplementation | 30 minutes before and 30 minutes after exercise completion at baseline and after 8 weeks of supplementation.
  Total Antioxidant Status (TAS) in serum will be measured to gauge overall antioxidant capacity. Higher levels indicate a stronger antioxidant defense.
Change from Baseline in Serum Superoxide Dismutase Activity 30 Minutes Before and 30 Minutes After Exercise Completion at 0 and 8 Weeks of Supplementation | 30 minutes before and 30 minutes after exercise completion at baseline and after 8 weeks of supplementation.
  Serum superoxide dismutase (SOD) activity, an antioxidant enzyme, will be measured to assess the body's defense against superoxide radicals. Higher activity levels indicate greater antioxidative defense.
Change from Baseline in Serum Protein Carbonyl Levels 30 Minutes Before and 30 Minutes After Exercise Completion at 0 and 8 Weeks of Supplementation | 30 minutes before and 30 minutes after exercise completion at baseline and after 8 weeks of supplementation.
  Serum protein carbonyls, markers of oxidative damage to proteins, will be measured. Higher levels indicate increased protein oxidation and cellular stress.
Change from Baseline in Serum Uric Acid Levels 30 Minutes Before Exercise at 0 and 8 Weeks of Supplementation | 30 minutes before exercise at baseline and after 8 weeks of supplementation.
  Serum uric acid will be measured as an indicator of purine metabolism and antioxidant activity, where higher levels may indicate greater antioxidant activity or metabolic changes.
Change from Baseline in Serum IgA Levels 30 Minutes Before Exercise at 0 and 8 Weeks of Supplementation | 30 minutes before exercise at baseline and after 8 weeks of supplementation.
  Immunoglobulin A (IgA) levels in serum will be measured to assess immune function, with higher levels indicating a robust immune response
Change from Baseline in Serum IgM Levels 30 Minutes Before Exercise at 0 and 8 Weeks of Supplementation | 30 minutes before exercise at baseline and after 8 weeks of supplementation.
  Immunoglobulin M (IgM) levels in serum will be measured to assess immune function, with higher levels indicating a robust immune response
Change from Baseline in Serum IgG Levels 30 Minutes Before Exercise at 0 and 8 Weeks of Supplementation | 30 minutes before exercise at baseline and after 8 weeks of supplementation.
  Immunoglobulin G (IgG) levels in serum will be measured to assess immune function, with higher levels indicating a robust immune response
Change from Baseline in Serum Creatine Kinase Levels 30 Minutes Before and 30 Minutes After Exercise Completion at 0 and 8 Weeks of Supplementation | 30 minutes before and 30 minutes after exercise completion at baseline and after 8 weeks of supplementation.
  Serum creatine kinase (CK), a marker of muscle damage, will be measured. Higher CK levels indicate greater muscle stress or damage.
Change from Baseline in Perceived Soreness (DOMS) Using Visual Analog Scale (VAS) at 30 Minutes Before and 30 Minutes After Exercise Completion at 0 and 8 Weeks of Supplementation | 30 minutes before and 30 minutes after exercise completion at baseline and after 8 weeks of supplementation.
  Delayed onset muscle soreness (DOMS) will be self-rated using a 10-point visual analog scale (VAS), where 0 indicates no soreness and 10 represents extreme soreness.
Change from Baseline in Perceived Recovery Using Visual Analog Scale (VAS) at 30 Minutes Before and 30 Minutes After Exercise Completion at 0 and 8 Weeks of Supplementation | 30 minutes before and 30 minutes after exercise completion at baseline and after 8 weeks of supplementation.
  Recovery will be self-rated by participants on a 10-point VAS, where 0 represents no recovery and 10 represents full recovery.
Change from Baseline in Perceived Soreness (DOMS) of Quadriceps Using a Digital Algometer 30 Minutes Before and 30 Minutes After Exercise Completion at 0 and 8 Weeks of Supplementation | Approximately 30 minutes before and 30 minutes after exercise completion at baseline (0 weeks) and after 8 weeks of supplementation.
  Perceived muscle soreness in the quadriceps will be assessed using a digital algometer, which applies consistent pressure to measure pain threshold and discomfort. Higher readings indicate higher resistance to soreness, while lower values indicate increased perceived soreness.
Daily Self-Report Diary on Upper Respiratory Tract and Gastrointestinal Symptoms Over 8 Weeks of Supplementation | Daily throughout the 8-week supplementation period.
  Participants will complete a daily diary to self-report any symptoms related to upper respiratory tract infections (URTI) and gastrointestinal (GI) health throughout the 8-week supplementation period. This diary will track symptom type, severity, and duration.
Change from Baseline in Gastrointestinal Symptoms Using the Gastrointestinal Symptom Rating Scale (GSRS) Before and After 8 Weeks of Supplementation | Baseline (pre-supplementation) and after 8 weeks of supplementation.
  The Gastrointestinal Symptoms Rating Scale (GSRS) will assess GI symptoms across multiple dimensions, including abdominal pain, reflux, indigestion, diarrhea, and constipation. Scores range from 1 (no discomfort) to 7 (severe discomfort) on each dimension, with higher scores indicating greater symptom severity.
Change from Baseline in Generalized Anxiety Disorder-7 (GAD-7) Score Before and After 8 Weeks of Supplementation | Baseline (pre-supplementation) and after 8 weeks of supplementation
  The GAD-7, a 7-item self-report questionnaire, will assess anxiety levels. Scores range from 0 to 21, with higher scores indicating greater anxiety severity. The questionnaire will be completed by participants before and after supplementation.
Change from Baseline in Perceived Restfulness Using Visual Analog Scale (VAS) After 0 and 8 Weeks of Supplementation | After 0 and 8 weeks of supplementation.
  Perceived restfulness will be assessed using a 10-point Visual Analog Scale (VAS), where 0 represents no restfulness and 10 represents feeling fully rested. Participants will complete the scale at baseline and at the end of the supplementation period.
Change from Baseline in Perceived Sleep Quality Using Visual Analog Scale (VAS) After 0 and 8 Weeks of Supplementation | After 0 and 8 weeks of supplementation.
  Perceived sleep quality will be rated on a 10-point Visual Analog Scale (VAS), with 0 indicating poor sleep quality and 10 indicating excellent sleep quality. Participants will complete the scale at baseline and after the supplementation period.
Change from Baseline in Pittsburgh Sleep Quality Index (PSQI) Score Before and After 8 Weeks of Supplementation | Baseline (pre-supplementation) and after 8 weeks of supplementation.
  The Pittsburgh Sleep Quality Index (PSQI), a self-rated questionnaire, assesses overall sleep quality and disturbances over a 1-month period. Scores range from 0 to 21, with higher scores indicating worse sleep quality. The PSQI will be completed at baseline and after the supplementation period.
Change from Baseline in Running Distance (Miles) Covered During 10-Minute Time Trial After 0 and 8 Weeks of Supplementation | After 0 weeks (baseline) and after 8 weeks of supplementation.
  The total distance in miles covered during a 10-minute running time trial will be measured to assess exercise performance. Greater distance covered indicates improved aerobic capacity and endurance.
Change from Baseline in Heart Rate (bpm) During Treadmill Running at 70-75% VO2Peak Assessed at 0, 15, 30, and 45 Minutes After 0 and 8 Weeks of Supplementation | 0, 15, 30, and 45 minutes during treadmill running at baseline (0 weeks) and after 8 weeks of supplementation.
  Heart rate, measured in beats per minute (bpm), will be assessed throughout treadmill running to monitor cardiovascular response. Lower heart rates at a set intensity indicate improved cardiovascular efficiency.
Change from Baseline in Rating of Perceived Exertion (RPE) During Treadmill Running at 70-75% VO2Peak Assessed at 0, 15, 30, and 45 Minutes After 0 and 8 Weeks of Supplementation | 0, 15, 30, and 45 minutes during treadmill running at baseline (0 weeks) and after 8 weeks of supplementation.
  RPE will be recorded using the Borg scale (6-20), where higher values indicate greater perceived effort. Lower RPE values at a fixed intensity suggest improved endurance and perceived ease of exercise.
Change from Baseline in Blood Lactate Levels (mmol/L) During Treadmill Running at 70-75% VO2Peak Assessed at 0, 15, 30, and 45 Minutes After 0 and 8 Weeks of Supplementation | 0, 15, 30, and 45 minutes during treadmill running at baseline (0 weeks) and after 8 weeks of supplementation.
  Blood lactate, measured in mmol/L, will be assessed as a marker of metabolic stress, with lower levels indicating improved lactate clearance and aerobic efficiency.
Change from Baseline in Blood Glucose Levels (mg/dL) During Treadmill Running at 70-75% VO2Peak Assessed at 0, 15, 30, and 45 Minutes After 0 and 8 Weeks of Supplementation | 0, 15, 30, and 45 minutes during treadmill running at baseline (0 weeks) and after 8 weeks of supplementation.
  Blood glucose, measured in mg/dL, will be monitored to assess energy utilization. Stable or lower levels may indicate improved metabolic flexibility.
Change from Baseline in Fat Oxidation Rate (g/min) During Treadmill Running at 70-75% VO2Peak Assessed at 0, 15, 30, and 45 Minutes After 0 and 8 Weeks of Supplementation | 0, 15, 30, and 45 minutes during treadmill running at baseline (0 weeks) and after 8 weeks of supplementation.
  Fat oxidation rate, measured in grams per minute (g/min), will be assessed to evaluate substrate utilization, with higher rates suggesting greater reliance on fat as an energy source.
Change from Baseline in Carbohydrate Oxidation Rate (g/min) During Treadmill Running at 70-75% VO2Peak Assessed at 0, 15, 30, and 45 Minutes After 0 and 8 Weeks of Supplementation | 0, 15, 30, and 45 minutes during treadmill running at baseline (0 weeks) and after 8 weeks of supplementation.
  Carbohydrate oxidation rate, measured in grams per minute (g/min), will be assessed to evaluate energy source utilization, with lower rates indicating improved fat utilization at moderate intensities.
Daily Self-Reported Adverse Event (AE) Log Throughout 8-Week Supplementation Period | Daily throughout the 8-week supplementation period.
  Participants will complete a daily self-report diary to record any adverse events (AEs) experienced, detailing the type, severity, duration, and any related symptoms. This log will help monitor the safety and tolerability of the supplementation over the study period.

OTHER OUTCOMES:
Change from Baseline in Gut Microbiome Composition Using Shotgun Metagenomic Sequencing (Fecal) During the 24 Hours Before and 24 Hours After Exercise Completion at 0 and 8 Weeks of Supplementation | 24 hours before and 24 hours after exercise completion at baseline (0 weeks) and after 8 weeks of supplementation.
  Shotgun metagenomic sequencing will analyze the composition and diversity of the gut microbiome in fecal samples. This measure provides insights into microbiome changes related to supplementation and exercise, with results expressed as relative abundance and diversity of microbial species.
Change from Baseline in Fecal Metabolomic Profile During the 24 Hours Before and 24 Hours After Exercise Completion at 0 and 8 Weeks of Supplementation | 24 hours before and 24 hours after exercise completion at baseline (0 weeks) and after 8 weeks of supplementation.
  Fecal metabolomic analysis will assess the profile of metabolites produced by the gut microbiota, providing insights into metabolic changes. Metabolite concentrations will be reported, with changes potentially reflecting shifts in gut microbial activity and metabolic byproducts.

CONTACTS AND LOCATIONS:
Overall Officials: Chad M Kerksick, PhD, Principal Investigator — Lindenwood University
Locations (1):
- Exercise and Performance Nutrition Laboratory, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.